CLINICAL TRIAL: NCT00606190
Title: Prospective Randomized Study of Brain Protection During Aortic Arch Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5985 Aortic Arch
Record Dates: First submitted 2007-12-27; First posted 2008-02-01 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Aneurysm of Aortic Arch
MeSH Terms: conditions — Aneurysm, Aortic Arch

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Retrograde brain perfusion (Active Comparator): Pt may be randomized to retrograde brain perfusion when having a repair of the ascending aortic artery (aorta) including the aortic arch. This is one of the standard methods used while the body and the brain are cooled down to sub-normal levels (hypothermia). This will take place while on the heart-lung machine.
  Interventions: Procedure: Retrograde brain perfusion
- Antegrade brain perfusion (Active Comparator): Pt may be randomized to antegrade brain perfusion when having a repair of the ascending aortic artery (aorta) including the aortic arch. This is one of the standard methods used while the body and the brain are cooled down to sub-normal levels (hypothermia). This will take place while on the heart-lung machine.
  Interventions: Procedure: Antegrade brain perfusion

INTERVENTIONS:
Procedure: Retrograde brain perfusion — observational
  Arms: Retrograde brain perfusion
Procedure: Antegrade brain perfusion — observational
  Arms: Antegrade brain perfusion

SUMMARY:
The purpose of this research study is to evaluate two standard approaches of supplying blood and oxygen to your brain during open heart surgery.

DETAILED DESCRIPTION:
The purpose of the clinical trial is to assess the best method of protecting the brain during long periods of circulatory arrest. The significance of this project will be to determine which method of brain protection (1) retrograde brain perfusion or (2) perfusion of the right subclavian artery with antegrade perfusion of the brain protects against brain injury after total arch replacement. Thus reducing the risk of stroke or neurocognitive deficits in patients undergoing this critical surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing a total arch replacement
* Less than 75 years old

Exclusion Criteria:

* EF less than 35%
* Pt shows evidence of major illness e.g. severe hepatic disease, severe renal failure, active cancer or major infection
* Pt unable to complete preop neuro assessment
* Pt is unwilling or able to complete followup requirements
* Pt is already enrolled in other new device or drug protocols that have not completed the primary endpoint or that clinically interferes with study endpoint
* Pt is a female who is pregnant or lactating
* Pt has history of stroke

Ages: 21 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2003-06; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
To determine what is the best method of brain protection during long periods of circulatory arrest | 6 months

SECONDARY OUTCOMES:
Will one method of brain protection be better than the other in prevention of post-op stroke and which method will provide freedom from postop neurobehavioural deficit at 6 months postop. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lars Svensson, MD, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Svensson LG, Blackstone EH, Apperson-Hansen C, Ruggieri PM, Ainkaran P, Naugle RI, Lima B, Roselli EE, Cooper M, Somogyi D, Tuzcu EM, Kapadia S, Clair DG, Sabik JF 3rd, Lytle BW. Implications from neurologic assessment of brain protection for total arch replacement from a randomized trial. J Thorac Cardiovasc Surg. 2015 Nov;150(5):1140-7.e11. doi: 10.1016/j.jtcvs.2015.07.054. Epub 2015 Jul 26. PMID 26409997